CLINICAL TRIAL: NCT06939309
Title: Efficacy of Acupuncture for Shoulder Pain Based on Remote Point Selection According to the Meridians
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH113-REC3-192
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Shoulder Pain; Acupuncture; Meridians
Keywords: Shoulder pain; Acupuncture; Meridians
MeSH Terms: conditions — Shoulder Pain | interventions — Acupuncture Therapy; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture SC Group (Experimental): The most affected meridian is determined based on location and movements. The physician first applies acupuncture to one standardized acupoint (LI10, TE7, SI7, or LU6) on the most affected meridian. After 3 minutes (3 minutes after the first acupuncture), the assessor performs the first evaluation. The physician then applies acupuncture to a controlled acupoint (PC6) not directly related to shoulder function. After another 5 minutes (8 minutes after the first acupuncture), the assessor performs the second evaluation. The final evaluation is conducted 30 minutes after the first acupuncture. The patient is instructed to perform shoulder movements throughout the treatment.
  Interventions: Procedure: Acupuncture
- Acupuncture CS Group (Experimental): The most affected meridian is determined using the same method by location and movements. The physician first applies acupuncture to the controlled acupoint (PC6). After 3 minutes, the assessor performs the first evaluation. The physician then applies acupuncture to one standardized acupoint (LI10, TE7, SI7, or LU6) on the most affected meridian. After another 5 minutes (8 minutes after the first acupuncture), the assessor performs the second evaluation. The final evaluation is conducted 30 minutes after the first acupuncture. The patient is instructed to perform shoulder movements throughout the treatment.
  Interventions: Procedure: Acupuncture
- Rehabilitation Group (Active Comparator): Participants will complete a 30-minute rehabilitation session, followed by an outcome assessment.
  Interventions: Procedure: Rehabilitation

INTERVENTIONS:
Procedure: Acupuncture — In this study, both the acupuncture SC group and the acupuncture CS group will receive two acupuncture treatments in one session. The SC group will first receive acupuncture at the standardized acupoint followed by the controlled acupoint, while the CS group will first receive acupuncture at the controlled acupoint followed by the standardized acupoint.
  Arms: Acupuncture CS Group; Acupuncture SC Group
Procedure: Rehabilitation — Participants will complete a 30-minute rehabilitation session, which includes electrotherapy and thermotherapy applied to the shoulder.
  Arms: Rehabilitation Group

SUMMARY:
This double blind randomized controlled trial investigates the immediate efficacy of acupuncture for shoulder pain using remote point selection based on meridian theory. A total of 90 participants with shoulder pain (Numerical Rating Scale ≥ 4) will be randomly assigned in a 1:1:1 ratio to one of three groups: acupuncture SC, acupuncture CS, and rehabilitation. Meridian selection will be determined based on the patient's most painful shoulder movement and corresponding pain location, followed by standardized distal acupoint application. Outcome measures include changes in pain intensity (NRS) and shoulder range of motion assessed at baseline, post-first acupuncture, post-second acupuncture, and 30 minutes post-treatment. Blinded evaluators will conduct all assessments. The study aims to assess the effectiveness of meridian-based remote acupuncture and explore its relationship with shoulder movement patterns and soft tissue involvement.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old.
* Shoulder pain persisting for at least one week.
* Numerical Rating Scale (NRS) score ≥ 4.

Exclusion Criteria:

* Patients with cervical radiculopathy or other localized neurological disorders affecting the upper limb.
* Psychiatric disorders that may interfere with examination, treatment, or evaluation of disease progression.
* Pregnant patients.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-18 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Numerical Rating Scale, NRS: 0-10) | Baseline evaluation before intervention. First evaluation: 3 minutes after the first acupuncture. Second evaluation: 3 minutes after the second acupuncture (8 minutes after the first). Final evaluation: 30 minutes after the first acupuncture.
  Patients will be asked to rate their pain intensity using a numerical scale. 0: No pain. 1-3: Mild pain - the patient feels pain but can tolerate it; normal daily activities and sleep are not disturbed.
  4-6: Moderate pain - the pain is noticeable and difficult to tolerate; sleep may be disturbed, such as waking up due to pain; patients may request pain medication.
  7-10: Severe pain - the pain is intense and intolerable; sleep is severely disturbed or impossible; pain medication is often necessary.

SECONDARY OUTCOMES:
Range of Motion | Baseline evaluation before intervention. First evaluation: 3 minutes after the first acupuncture. Second evaluation: 3 minutes after the second acupuncture (8 minutes after the first). Final evaluation: 30 minutes after the first acupuncture.
  A goniometer will be used to measure the range of motion of the affected shoulder joint in the following movements: flexion, abduction, external rotation, and internal rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Hospital, Ministry of Health and Welfare, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policy and data privacy considerations. The study data include sensitive health information that cannot be fully de-identified, and there are currently no resources allocated for managing data sharing requests.

REFERENCES:
- [Result] Chandran KP, Chandran PP, Arumugam N, Muthappan S. Effect of Remote and Local Acupuncture Points on Periarthritis of Shoulder: A Comparative Study. J Acupunct Meridian Stud. 2021 Feb 28;14(1):13-20. doi: 10.51507/j.jams.2021.14.1.13. PMID 35770597
- [Result] Chen IW, Liao YT, Tseng H, Lin HC, Chou LW. Pain, function and peritendinous effusion improvement after dry needling in patients with long head of biceps brachii tendinopathy: a single-blind randomized clinical trial. Ann Med. 2024 Dec;56(1):2391528. doi: 10.1080/07853890.2024.2391528. Epub 2024 Aug 14. PMID 39140690
- [Result] Takakura N, Takayama M, Kawase A, Kaptchuk TJ, Kong J, Vangel M, Yajima H. Acupuncture for Japanese Katakori (Chronic Neck Pain): A Randomized Placebo-Controlled Double-Blind Study. Medicina (Kaunas). 2023 Dec 9;59(12):2141. doi: 10.3390/medicina59122141. PMID 38138244
- [Result] Calamita SAP, Biasotto-Gonzalez DA, De Melo NC, Fumagalli MA, Amorim CF, de Paula Gomes CAF, Politti F. Immediate Effect of Acupuncture on Electromyographic Activity of the Upper Trapezius Muscle and Pain in Patients With Nonspecific Neck Pain: A Randomized, Single-Blinded, Sham-Controlled, Crossover Study. J Manipulative Physiol Ther. 2018 Mar-Apr;41(3):208-217. doi: 10.1016/j.jmpt.2017.09.006. PMID 29549891
- [Result] Ben-Arie E, Kao PY, Lee YC, Ho WC, Chou LW, Liu HP. The Effectiveness of Acupuncture in the Treatment of Frozen Shoulder: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2020 Sep 25;2020:9790470. doi: 10.1155/2020/9790470. eCollection 2020. PMID 33062030
- [Result] Green S, Buchbinder R, Hetrick S. Acupuncture for shoulder pain. Cochrane Database Syst Rev. 2005 Apr 18;2005(2):CD005319. doi: 10.1002/14651858.CD005319. PMID 15846753
- [Result] Schroder S, Meyer-Hamme G, Friedemann T, Kirch S, Hauck M, Plaetke R, Friedrichs S, Gulati A, Briem D. Immediate Pain Relief in Adhesive Capsulitis by Acupuncture-A Randomized Controlled Double-Blinded Study. Pain Med. 2017 Nov 1;18(11):2235-2247. doi: 10.1093/pm/pnx052. PMID 28371868